CLINICAL TRIAL: NCT07024108
Title: Comparison Between Perfusion Index and Pulse Pressure Variability for Prediction of Intravascular Volume During Major Abdominal Surgeries
Status: Active, not recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MS 73/2025
Record Dates: First submitted 2025-04-26; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-02

CONDITIONS: Comparison Between Perfusion Index and Pulse Pressure Variability for Prediction of Intravascular Volume During Major Abdominal Surgeries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Each year, at least 310 million patients undergo major surgery worldwide, procedures that involve the administration of intravenous fluids Intraoperative hemodynamic management is challenging because precise assessment of the adequacy of the intravascular volume is difficult during surgery Achieving optimal IV fluid therapy should improve perioperative outcomes and is a key component in many perioperative guidelines and pathways. IV fluids, like other medications, should only be given in well-defined protocols according to individual needs More recently, so called dynamic predictors of fluid responsiveness such as pulse pressure variation (PPV), stroke volume variation (SVV), or Perfusion Index (PI) have been used in intraoperative goal directed fluid therapy ( GDT) hemodynamic protocols

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

ASA 1, 2 Age: 18-65 Undergoing major abdominal surgeries Mechanically ventilated and sedated patients

Exclusion Criteria:

Chronic cardiac arrhythmias High doses of vasopressors Altered myocardial function (left ventricular ejection fraction < 50%) Peripheral vascular disease Severe respiratory disease Pulmonary or intra-abdominal hypertension Open chest

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adult patients under general anaesthesia scheduled for major abdominal surgeries between the period from January 2025 to june 2025 will be observed for comparison between PI and PPV in detecting intravascular volume.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-08-03 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Comparison between perfusion index and pulse pressure variability for prediction of intravascular volume during major abdominal surgeries | 6 months
  Comparing 2 percentage; Perfusion index and pulse pressure variability in assessment of intravascular volume and fluid responsiveness of the patient during major abdominal surgeries PI is a ratio of pulsatile light absorption to continuous light absorption, denoted as AC/DC.
  Normal PI values can vary widely, ranging from less than 1% to greater than 10%.
  The pulse pressure variation (PPV) is a percentage measure of the respiratory effect on the variation of systemic arterial blood pressure in patients receiving full mechanical ventilation The PI will be monitored by attaching a sensor to the patient's finger (Ultralife Pulse Oximeter JPD-500D).
  The PPV will be measured using an arterial line in radial artery Patients will receive maintenance and deficit fluids then measuring perfusion index (PI) and pulse pressure variability (PPV) which the cut off value of is higher than 13% for more than 5 min, values of PI in percentage in corresponding time will be measured and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Randa Ali Shokry, Study Chair — Faculty of medicine AinShamsU
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt